CLINICAL TRIAL: NCT00989131
Title: An Open, Randomized, Multicenter Study in Patients With Recurrent Epithelian Cancer, Primary Peritoneal Cancer or Fallopian Tube Cancer to Compare the Efficay and Safety of Paclitaxel (Micellar) Nanoparticles and Paclitaxel (Cremophor® EL)
Brief Title: Study of Paclitaxel in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oasmia Pharmaceutical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OAS-07OVA
Record Dates: First submitted 2009-09-28; First posted 2009-10-02 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel, micellar (Paclical®) (Experimental)
  Interventions: Drug: Paclical®
- Paclitaxel, CrEL (Taxol®) (Active Comparator)
  Interventions: Drug: Taxol®

INTERVENTIONS:
Drug: Paclical® — 250 mg/m2 of Paclical® is given as a one-hour IV infusion, followed by carboplatin, on day 1 of each 21 day cycle.
  Number of Cycles: 6. Cycle 2-6 will be given with 3 weeks interval between treatments.
  Arms: Paclitaxel, micellar (Paclical®)
Drug: Taxol® — 175 mg/m2 of Taxol® is given as 3 hour IV infusion, followed by carboplatin on day 1 of each 21 day cycle.
  Number of Cycles: 6. Cycle 2-6 will be given with 3 weeks interval between treatments.
  Arms: Paclitaxel, CrEL (Taxol®)

SUMMARY:
RATIONALE: Paclitaxel is one of the most widely used human anticancer agents. Paclitaxel has a low degree of solubility and Cremophor EL is typically used as the solubiliser. Cremophor EL is known to cause hypersensitivity reactions that can be life-threatening. As Paclical® does not contain Cremophor EL, hypersensitivity reactions can be expected to be less.

PURPOSE: To study the efficay and safety of two different formulations of paclitaxel, Paclical® and Taxol®.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer.
* Patients relapsing > 6 months after end of first line or second line treatment including platinum based therapy. Prior therapy and duration of response will be documented in the CRF for descriptive analysis.
* CA 125 >2 x upper normal limit (UNL) documented at two occasions, with more than one week interval, according to appendix I, patient groups A and B, measurable/non- measurable disease.
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) performance score 0-2
* Life expectancy >12 weeks
* Patient has blood counts at baseline of:

  * Absolute neutrophil count (ANC) >1,5 x 109 / L.
  * Platelet count >100 x 109 / L
  * Haemoglobin (Hb) ≥9g/dl (can be post transfusion)
* Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) < 2 x UNL
* Total bilirubin ≤1.5 x UNL.
* Adequate renal function defined as serum creatinine < 2.0 mg/dl or 177μmol/l.
* Alkaline phosphatase (ALP) < 2.5 x UNL
* Signed informed consent obtained

Exclusion Criteria:

* Patient has peripheral neuropathy of grade ≥ 2 per NCI-CTCAE version 3.0
* Surgical procedure due to progressive disease within 4 weeks of any of the CA-125 measurements
* Patient receiving concurrent hormonal, immuno-, or radiotherapy. Treatment must have stopped for at least 4 weeks before start of drug treatment (Day 1, Cycle 1).
* Bowel obstruction at screening
* Tumours of other origin or histology
* Patient of child-bearing potential, not practising adequate contraception, or pregnant or lactating women
* Patient has a history of severe allergy or severe hypersensitivity to study drugs
* Any uncontrolled medical problem that in the opinion of the investigator would preclude safe administration of the study drugs, e.g. heart, lung or kidney disease, suspicion of brain metastasis or mental disorder to make the patient unable to participate in the study
* Participation in an investigational drug study within 4 weeks prior to study treatment (Day 1, Cycle 1)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2009-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS).
Change in Area under the curve of CA 125
Incidence and severity of hypersensitivity reactions

SECONDARY OUTCOMES:
Nadir and time to nadir of CA 125 during and after treatment
T½ of CA 125
Safety and tolerability
Response rate using CA 125
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ignace Vergote, Prof., Principal Investigator — Division of Gynaecological Oncology, Department of Obstetrics and Gynaecology, University Hospitals Leuven, Belgium
Locations (84):
- Belarus (4):
  - Gomel Regional Clincial Oncology Center, Homyel
  - Minsk City Clinical Oncology Hospital, Minsk
  - Alexandrov National Cancer Center of Belarus, Minsk
  - Vitebsk Regional Clinical Oncology Center, Vitebsk
- Department of gyneacology, Campus Gasthuisberg, Leuven, Belgium
- Bulgaria (3):
  - Regional Oncology Dispensary, Shumen
  - Hospital for a Active Treatment, Tsaritsa Yoanna, Sofia
  - Regional Oncology Dispensary, Stara Zagora
- Croatia (3):
  - Klinički Bolnički Centar Rijeka, Rijeka
  - Klinički Bolnički Centar Split, Split
  - Klinikčki Bolnički Centar Zagreb, Zagreb
- Czechia (4):
  - Onkologická klinika, Fakultní nemocnice Královské Vinohrady, Olomouc
  - Onkologické a radioterapeutické oddělení, Fakultní nemocnice Plzeň, Pilsen
  - Radioterapeutická a onkologická klinika, Fakultní nemocnice Královské Vinohrady, Prague
  - Ústav radiační onkologie, Fakultní nemocnice Na Bulovce, Prague
- Onkologisk Afdelning, Herning Sygehus, Herning, Denmark
- Finland (2):
  - Kuopion Yliopistollinen Sairaala, Naisten Klinikka, Kuopio
  - Turun Yliopistollinen Keskussairaala, Naisten Klinikka,, Turku
- Hungary (5):
  - Kaposi Mór Megyei Kórház, Onkológiai Tanszék, Kaposvár
  - B.-A.-Z. Megyei Kórház és Egyetemi Oktató Kórház, Észak-Kelet Magyarországi Regionális Klinikai Farmakológiai Központ, Miskolc
  - Szabolcs-Szatmár-Bereg Megyei Önkormányzat Jósa András Oktató Kórháza, Onkoradiológia, Nyíregyháza
  - Veszprém Megyei Csolnoky Ferenc Kórház-Rendelőintézet ZRT, Veszprém
  - Zala Megyei Kórház, Onkológia, Zalaegerszeg
- Latvian Oncology Center of Riga Easter Hospital Ltd, Riga, Latvia
- Lithuania (2):
  - Kaunas Medical University Hospital, Oncology Clinic, Kaunas
  - Institute of Oncology, Vilnius University, Vilnius
- Romania (4):
  - County Clinical Emergency Hospital Oradea, Oradea, Bihor County
  - MEDITECH SRL, ORIZONT Polyclinic, Craiova, Dolj
  - Cluj CF University Hospital, Cluj-Napoca
  - Constanta Clinical County Hospital, Constanța
- Russia (26):
  - State Institution, Moscow City Oncology Hospital #62, Moscow, Krasnogorsky Region
  - State Medical Institution "Stavropol Regional Clinical Oncology Center", Stavropol, Stavropol Kray
  - State Medical Institution, Arkhankelsk Regional Clinical Oncology Center, Arkhangelsk
  - State Medical Institution, Altai Regional Oncology Center, Barnaul
  - Chelyabinsk Regional Clinical Oncology Center, Chelyabinsk
  - Clinical Oncology Center, Kazan'
  - State Treatment and Prevention Institution, Kirov Regional Clinical Oncology Center, Kirov
  - State Medical Institution "Clinical Oncology Center #1" under the Ministry of Health of Krasnodar Region, Krasnodar
  - State Medical Institution, Regional Oncology Center #2, Surgery department, Magnitogorsk
  - N.N. Blokhin Cancere Research Center under the Russian Academy of Medical Sciences, Moscow
  - Federal State Institution, Central Clinical Hospital with Outpatient Unit under the Russian Presidential Administration, Moscow
  - Federal State Institution "Privolzhskiy District Medical Center of Federal Bio-medical Agency", Nizhny Novgorod
  - State Medical Institution of the Omsk Region, Clincial Oncology center, Omsk
  - State Medical Institution "Orenburg Regional Clinical Oncology Center", Orenburg
  - State Medicinal Institution, Reginal oncology center, Penza
  - State Medical Institution "Republic Oncology Center", Petrozavodsk
  - Pyatigorsk Affiliate of State Medical Institution, Stavropol Regional Clinical Oncology Center, Pyatigorsk
  - State Medical Institution "Leningrad Regional Oncology Center", Saint Petersburg
  - Federal State Medical Institution, N.N. Petrov Research Institute of Oncology under the Federal Agency for High-Tech Medical Care of the Russian Federation, Oncogynecology Department, Saint Petersburg
  - St Petersburg State Medical Institution, City clinical oncology center, Saint Petersburg
  - Samara Regional Clinical Oncology Center, Samara
  - State Medical Institution, Oncology Center #2 under the Krasnodar Region Healthcare Department, Sochi
  - State Medical Institution, Tambov Regional Oncology Center #2, Tambov
  - State Medical Institution, Voronezh Regional Clinical Oncology Center, Voronezh
  - State Medical Institution of the Yaroslavl, Region Clinical Oncology Center, Yaroslavl
  - State Budget-funded Medical Institution of Sverdlovsk Region "Sverdlovsk Regional Oncology Center", Yekaterinburg
- Serbia (4):
  - Institut za onkologiju i radiologiju Srbije, Klinika za medikalnu onkologiju, Belgrade
  - Institut za onkologiju Vojvodine, Klinika za operativnu onkologiju, Kamenitz
  - Klinički Bolnički Centar Kragujevac, Centar za onkologiju i radioterapiju, Kragujevac
  - Klinički Centar Niš, Klinika za onkologiju, Niš
- Slovakia (3):
  - Onkologicke oddelenie, FNsP F. D. Roosevelta, Banska Bysterica
  - Interne oddelenie, Narodny onkologicky ustav, Bratilslava
  - Crimean Republicann Oncology Dispensary, Simferopol
- Sweden (5):
  - Divisionen för Onkologi , Sahlgrenska Universitetssjukhuset, Gothenburg
  - Onkologikliniken, Universitetssjukhuset Linköping, Linköping
  - Onkologiska Kliniken, Universitetssjukhuset Lund, Lund
  - Kliniken för Gynekologisk Onkologi, Regionsjukhuset, Örebro
  - Gyn-Onkologiska kliniken, Norrlands universitetssjukhus, Umeå
- Ukraine (16):
  - Kyiv Regional Oncology Center, Kyiv, Bagautivska Str. 1
  - Kharkiv Regional Clinical Oncology, Kharkiv, Lisoparkivska Str 4
  - Ivano-Frankivsk Regional Oncology Center, Ivano-Frankivsk, Medychna Str.17
  - Cherkassy Regional Oncological Centre, Cherkassy
  - Cherkassy Regional Oncological Centre, Chernivtsy
  - KZ, City Clinical Hospital #19 City oncology Center, Dnipro
  - Multi-profile clinical hospital#4, Dnipropetrovsk
  - Donetsk Regional Antitumor Center, Donetsk
  - "S.P. Grygoryev Institute of Medical Radiology of the Academy of Medical Science of Ukraine, Kharkiv
  - Kherson Reginal Oncological Center, Kherson
  - DU, National Institute of Cancer, Department of Oncogynecology, Kiev
  - Kiev City Oncology center, Kiev
  - Lugansk Regional Oncology Center, Luhansk
  - Odessa City Oncological Center, Odesa
  - Sumy Regional Onclolgy Center, Sumy
  - Ternopil Regional Oncology Hospital, Ternopil

REFERENCES:
- [Derived] Vergote I, Bergfeldt K, Franquet A, Lisyanskaya AS, Bjermo H, Heldring N, Buyse M, Brize A. A randomized phase III trial in patients with recurrent platinum sensitive ovarian cancer comparing efficacy and safety of paclitaxel micellar and Cremophor EL-paclitaxel. Gynecol Oncol. 2020 Feb;156(2):293-300. doi: 10.1016/j.ygyno.2019.11.034. Epub 2019 Dec 9. PMID 31826802